CLINICAL TRIAL: NCT04476719
Title: Open-Label, Randomised, Single Oral Dose, Two-Period, Cross-Over Trial To Assess The Bioequivalence Of Atafenovir 200 Mg Kapsul In Comparison With Arbidol 100 Mg Kapsul In Healthy Male Subjects Under Fasting Conditions
Brief Title: The Bioequivalence Study of Umifenovir 200 mg Capsul (ATABAY, Turkey) Under Fasting Conditions
Acronym: Umifenovir
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Atabay Kimya Sanayi Ticaret A.S. (Industry)
Collaborators: Novagenix Bioanalytical Drug R&D Center (Network); Farmagen Ar-Ge Biyot. Ltd. Sti (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NOV2020/01918
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-06

CONDITIONS: Bioequivalence
Keywords: COVID-19 drug treatment; Antiviral Agents; Umifenovir; Novagenix; Farmagen; Atabay
MeSH Terms: interventions — Drug Evaluation; umifenovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atafenovir 200 mg Kapsül (Experimental): Capsules containing 207.009 mg umifenovir hydrochloride monohydrate equivalent to 200 mg umifenovir hydrochloride (Atabay-Turkey).
  Interventions: Drug: ATAFENOVIR 200 MG KAPSUL
- Arbidol 100 mg Kapsül (Active Comparator): Capsules containing 103.504 umifenovir hydrochloride monohydrate equivalent to 100 mg umifenovir hydrochloride (OTC-Pharma Russia).
  Interventions: Drug: ARBIDOL 100 MG KAPSUL

INTERVENTIONS:
Drug: ATAFENOVIR 200 MG KAPSUL — A 200 mg capsule 0ral administration with 240 ml water
  Other Names: Test Drug
  Arms: Atafenovir 200 mg Kapsül
Drug: ARBIDOL 100 MG KAPSUL — Two 100 mg capsules will be administrated with 240 ml water orally.
  Other Names: Reference Drug
  Arms: Arbidol 100 mg Kapsül

SUMMARY:
A single dose of Reference product containing 200 mg umifenovir hydrochloride monohydrate equivalent to 200 mg umifenovir hydrochloride and a single dose of Test product containing 200 mg umifenovir hydrochloride monohydrate equivalent to 200 mg umifenovir hydrochloride or vice versa; administered with 240 mL of water at room temperature, in each period under fasting conditions with Covid-19 Pandemic precautions.

DETAILED DESCRIPTION:
In order to investigate the bioequivalence of all products, the 90% confidence intervals will be calculated for the geometric mean ratios of test and reference for Cmax and AUC0-tlast of umifenovir. These confidence intervals will then be compared with the corresponding acceptance ranges.

In order to achieve a better approximation to a normal distribution, Cmax and AUC0-tlast data for umifenovir will be logarithmically transformed (base e) before analysis. The sources of variation will be treatments, periods, sequences and subjects within the sequence. Evaluation of treatment, period, sequence and subject (nested within sequence) effects at 5% level of significance will be performed. From the result, the two one-sided hypothesis at the 5% level of significance will be tested by constructing the 90% confidence interval for the geometric mean ratios of test/reference products. The confidence interval is calculated by retransformation of the shortest confidence interval for the difference of the ln-transformed mean values. Differences in tmax will be evaluated non-parametrically.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian male subjects aged between 20 and 40 years,
2. Non smokers or smoking maximum 5 cigarettes a day, those who won't smoke or drink coffee during the study period,
3. Two Negative Covid-19 PCR test results.
4. Negative alcohol breath test results,
5. Normal physical examination at screening visit,
6. Having the Body Mass Index ranged between 18.5-30 kg/m2 (see Appendix I) which is in the desirable range according to the age,
7. Ability to communicate adequately with the investigator himself or his representatives,
8. Ability and agreement to comply with the study requirements,
9. Normal blood pressure and heart rate measured under stabilised conditions at the screening visit after at least 5 minutes of rest under supine position: SBP within 100 to 140 mmHg, DBP within 60 to 90 mmHg and HR within 50 to 90 bpm,
10. Normal/ acceptable 12-lead electrocardiographic results at least after 5 minutes of rest,
11. Laboratory results within normal range or clinically non-significant (CBC, glucose, urea, uric acid, creatinine, estimated GFR (eGFR), total bilirubin, sodium, potassium, calcium, chloride, SGOT (AST), SGPT (ALT), GGT, alkaline phosphatase, total protein and urinalysis), drug addiction scanning in urine results in negative (amphetamine, barbiturate, benzodiazepine, cannabinoid, cocaine, opiate),
12. Understanding of the study and agreement to give a written informed consent.

Exclusion Criteria:

1. Who have atopic constitution or asthma or known allergy for umifenovir and/or any other ingredients of the products.
2. Who have positive Covid-19 PCR test result.
3. Any history or presence of clinical relevance of cardiovascular, neurological, musculoskeletal, haematological, hepatic, gastrointestinal, renal, pulmonary, endocrinological, metabolism or psychiatric disease, any type of porphyria.
4. Symptomatic or asymptomatic orthostatic hypotension at screening or before the first drug administration defined by a decrease of SBP more than 20 mmHg or DBD more than 10 mmHg occurs between sitting/supine to standing position subject will be excluded (if it deemed necessary by the investigator),
5. Presence or history of malabsorption or any gastrointestinal surgery except appendectomy or except herniotomy.
6. Subjects who have given more than 400 mL blood within the last two months before the first drug administration and subjects who have participated to any drug research within the last two months before the first drug administration.
7. Subjects suspected to have a high probability of non-compliance to the study procedure and/or completion of the study according to the investigator's judgement.
8. Subjects who used any of prescribed systemic or topical medication (including OTC medication) within 2 weeks (or six elimination half lives of this medication, whichever is longer) before the initiation of the study (except single doses of analgesics which have no drug interaction with study product).
9. Use of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
10. History of allergic response to heparin.
11. Subjects who have any chronic disease which might interfere with absorption, distribution, metabolism or excretion of the drug.
12. Subjects who regular consumed of beverages or food containing methylxanthines (e.g. coffee, tea, cola, caffeine, chocolate, sodas,) equivalent to more than 500 mg methylxanthines per day.
13. Subjects who has taken any grapefruit or grapefruit juice during 7 days prior to drug administration, during the study.
14. History of drug abuse.
15. History of alcohol abuse and/or regular use of more than 2 units of alcohol per day or 10 units per week and/or positive alcohol breath test results (Note: one unit of alcohol equals 250 mL beer, 125 mL wine or 25 mL spirits).
16. Positive blood test for HBV, HCV and HIV.
17. Who have relationship to the investigator.
18. Who are not suitable to any of inclusion criteria.
19. History of difficulty of swallowing.
20. Intake of depot injectable solutions (including study medications) within 6 months before start of the study.
21. Intake of enzyme-inducing, organotoxic or long half-life drugs within 4 weeks before start of the study.
22. Special diet due to any reason, e.g. vegetarian.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-07-22 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
Primary PK Endpoint | 12 weeks
  AUC0-tlast umifenovir
Primary PK Endpoint | 13 weeks
  Cmax of umifenovir

SECONDARY OUTCOMES:
Secondary PK Endpoint | 14 weeks
  t1/2 of umifenovir
Secondary PK Endpoint | 15 weeks
  tmax of umifenovir
Secondary PK Endpoint | 16 weeks
  AUC0-inf of umifenovir

CONTACTS AND LOCATIONS:
Overall Officials: Muradiye Nacak, MD,PhD, Principal Investigator — Farmagen Ar-Ge Biyot. Ltd. Sti; Taner Ezgi, MD, Study Director — Farmagen Ar-Ge Biyot. Ltd. Sti
Locations (2):
- Turkey (Türkiye) (2):
  - Novagenix Drug R&D Center, Akyurt, Ankara
  - Farmagen Ar-Ge Biyot. Ltd. Sti., Şahinbey, Gaziantep